CLINICAL TRIAL: NCT05995197
Title: The Effect of Action Observation Therapy on Balance in Patients With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, melike özipek, physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedipolUmelikeözipek
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy; Exercise Therapy
Keywords: action observation therapy; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- action observation therapy group (Experimental): Children will watch the action observation therapy video on the computer screen placed 1 m in front of a chair in which they can sit comfortably, but they will not be allowed to move while watching the video. Children will watch the video of the exercise offered by the therapist and then practice the exercise. The watching time for each exercise is 3 minutes, and after watching 3 minutes, they will do the exercise in the video for 3 minutes.In order to increase the effectiveness of the action observation training. Children will be instructed to concentrate on the video at 1-minute intervals to allow children's attention span. The treatment program will be applied for 30 minutes, 5 days a week for 3 weeks. The first session of the exercise program will be held face-to-face and the other sessions will be followed online. Treatment will be started within the first 48 hours after the evaluation. After the applications, the evaluations at the beginning of the treatment will be repeated.
  Interventions: Other: action observation
- control group (No Intervention): Children with CP will watch the video on the computer screen placed 1 m in front of a chair in which they can sit comfortably, but they will not be allowed to move while watching the video. The therapist will explain the exercises verbally. Children will practice the exercise after watching cartoons. The watching time for each exercise is 3 minutes, and after watching 3 minutes of cartoons, they will do the exercise for 3 minutes. Children will be instructed to concentrate on the video at 1-minute intervals to allow children's attention span. The treatment program will be applied for 30 minutes, 5 days a week for 3 weeks. The first session of the exercise program will be held face-to-face and the other sessions will be followed online. Treatment will be started within the first 48 hours after the evaluation. After the applications, pre-treatment evaluations will be repeated.

INTERVENTIONS:
Other: action observation — cartoon observation
  Arms: action observation therapy group

SUMMARY:
type of study: clinical trial the goal of this study is to learn about action observation therapy for cerebral palsy population.

The main question it aim to answer is:

Is action observation therapy effective on balance in children with cerebral palsy? Twenty-four children who met the inclusion criteria in the study will be randomly divided into two groups as the training group(action observation group) and the control group.

DETAILED DESCRIPTION:
The history and demographic information of all cases will be obtained.Action observation therapy will be applied to improve balance. The therapist will verbally explain the program to be applied to both groups. Children with CP will watch the video on the computer screen placed 1 m in front of a chair in which they can sit comfortably, but they will not be allowed to move while watching the video. Children with CP will watch the video of the exercise offered by the therapist and then practice the exercise. The watching time for each exercise is 3 minutes, and after watching 3 minutes, they will do the exercise in the video for 3 minutes. The control group will be shown cartoons. After 3 minutes of monitoring, each exercise will be studied for 3 minutes. In order to increase the effectiveness of the action observation training, the participants will watch the video at the designated time in a quiet and noiseless place. Children will be instructed to concentrate on the video at 1-minute intervals to allow children's attention span. The treatment program will be applied for 30 minutes, 5 days a week for 3 weeks. The first session of the exercise program will be held face-to-face and the other sessions will be followed online. Treatment will be started within the first 48 hours after the evaluation. After the applications, the evaluations at the beginning of the session will be repeated.

Physiotherapy program to be applied:

First week:

* Double-leg balancing on soft ground with eyes open, hands free
* Balance on both feet on soft ground with eyes closed, hands free
* Stand on one leg with eyes open on hard ground
* Stand on one leg on hard ground with eyes closed

Second week:

* Standing with feet together on hard ground
* Standing in tandem on hard ground
* Right-left lower extremity weight transfer
* Step forward in standing position

Third week:

* Standing with feet together on soft ground
* Standing in tandem on soft ground
* Taking steps in different directions in a standing position
* Kicking the ball with the foot Pre- and post-treatment fNIRS imaging will be used to measure the cerebral cortex blood supply of the participants. The registration will be taken from the fNIRS device (Medical Technologies LLC, Berlin, Germany) using the program NIRStar Acquisition (NIRx Medizintechnik GmbH, Germany). Records will be taken to scan the bilateral supplementary motor area over 8 sources and 4 receivers. NIRS registration will take place during action observation therapy and balance tests. In measuring balance with action observation therapy; Resting in sitting position for 20 seconds, watching action observation video while sitting for 20 seconds, standing on two legs on hard ground for 20 seconds, resting in sitting position for 20 seconds, will be repeated 6 times. For evaluation on soft ground, 20 seconds of resting on both feet with eyes open, 20 seconds of watching action observation video, 20 seconds of standing on two feet with eyes open, 20 seconds of resting on both feet with eyes open will be applied and fNIRS measurement will be performed by repeating 6 times. The same periods will be applied to the control group and a cartoon will be watched instead of the action observation video.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with CP
* To be at I and II levels according to the Gross Motor Function Classification System
* Having bilateral and unilaterally affected spastic type CP
* Cooperating with assessments
* Absence of vision and hearing loss
* According to the health board report, only motor skills are affected

Exclusion Criteria:

* Botulinum toxin application in the last 6 months Having had any surgical operation in the last 6 months
* Having dyskinetic, ataxic and hypotonic type CP
* Not attending treatment sessions regularly for 2 weeks
* Not participating in the pre- and post-treatment evaluation

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric balance scale | 2 days before treatment and after 3 weeks
  The pediatric balance scale is a modified version of the Berg balance scale and is used to evaluate the functional balance ability of school-age children. The scale consists of 14 items, scored from 0 (lowest function) to 4 (highest function), with a maximum score of 56.

SECONDARY OUTCOMES:
Gross motor function classification system | 2 days before treatment
  The Gross Motor Function Classification System (KMFSS) for CP is based on self-initiated movements with an emphasis on sitting, displacement and mobility. The main criterion when defining the five-level classification system is that the differences between the levels are meaningful in everyday life.
  General titles of each level LEVEL I: Walks without restrictions. LEVEL II: Walks with restrictions. LEVEL III: Walks using hand-held mobility devices. LEVEL IV: Self-movement is limited. Can use a motorized mobility vehicle. LEVEL V: Transported in a manual wheelchair.
Gross motor function measurement-88 | 2 days before treatment and after 3 weeks
  Gross Motor Function Scale (GMFM-88) is divided into 5 main sections. It consists of a total of 88 items, 17 in the supine-prone position and turning section, 20 in the sitting section, 14 in the crawling-over-knee section, 13 in the standing section, and 24 in the walking-running-stair climbing section.
Lower Extremity Selective Control Evaluation Scale (SCALE) | 2 days before treatment and after 3 weeks
  The evaluation method currently used in the evaluation of selective motor control of the lower extremity is SCALE. Hip, knee, ankle, subtalar joint and toes bilaterally; It scores between 0-2 points.
Trunk Impairment Scale | 2 days before treatment and after 3 weeks
  The trunk impairment scale evaluates the trunk functionally in terms of strength in sitting position. The trunk impairment scale consists of three subsections: static, dynamic and coordination. The highest scores that can be obtained from the static, dynamic and coordination sub-headings are respectively; 7, 10 and 6 points. The total scale score ranges from 0 to 23.
Pediatric Outcome Data Collection Instrument (PODCI) | 2 days before treatment and after 3 weeks
  PODCI is one of the scales with proven validity and reliability, which is prepared for both children and adolescents, and is frequently used to determine functional status and evaluate health-related quality of life. The scale has 3 different forms;
  1. PODCI child form: The section consisting of 86 questions is filled by the families of children aged 6-10.
  2. PODCI adolescent family form: The section consisting of 86 questions is filled by the families of adolescents aged 11-18.
  3. PODCI adolescent form: The section consisting of 83 questions is filled by adolescents between the ages of 11-18.
  As a result, subscale standardized score "0" indicates worse health status and quality of life, "100" score indicates good health status and quality of life.
Nintendo Wii-Fit Balance Score | 2 days before treatment and after 3 weeks
  After the demographic information of the patient is saved in the device system, the patient is shown how to place his/her foot on the Nintendo Wii Fit balance board, the weight ratio given to the right and left feet (Body Center of Gravity right and left) is evaluated by asking him to stand on the balance board without moving, and the data is recorded as a percentage.
Timed Get Up and Go Test (TUG) | 2 days before treatment and after 3 weeks
  It is a valid and reliable method used to evaluate functional mobility and static and dynamic balance in CP. From a starting position with hips, knees, and ankles flexed to 90°, participants get up from a chair without arm support, walk 3 meters, return and sit in the chair. The time starts to be recorded with the "go" prompt given by the evaluator and is stopped when the hip touches the chair.
Functional Near Infrared Spectroscopy (fNIRS) Application | 2 days before treatment and after 3 weeks
  fNIRS is one of the new methods used in the measurement of local cerebral blood flow. It provides information about brain activity in the measured region using optical scattering and absorption of light at wavelengths close to infrared (700-950 nm).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abdelhaleem N, Taher S, Mahmoud M, Hendawy A, Hamed M, Mortada H, Magdy A, Raafat Ezz El-Din M, Zoukiem I, Elshennawy S. Effect of action observation therapy on motor function in children with cerebral palsy: a systematic review of randomized controlled trials with meta-analysis. Clin Rehabil. 2021 Jan;35(1):51-63. doi: 10.1177/0269215520954345. Epub 2020 Sep 9. PMID 32907374
- [Result] Jeong YA, Lee BH. Effect of Action Observation Training on Spasticity, Gross Motor Function, and Balance in Children with Diplegia Cerebral Palsy. Children (Basel). 2020 Jun 18;7(6):64. doi: 10.3390/children7060064. PMID 32570855
- [Result] Jung Y, Chung EJ, Chun HL, Lee BH. Effects of whole-body vibration combined with action observation on gross motor function, balance, and gait in children with spastic cerebral palsy: a preliminary study. J Exerc Rehabil. 2020 Jun 30;16(3):249-257. doi: 10.12965/jer.2040136.068. eCollection 2020 Jun. PMID 32724782
- [Result] Sgandurra G, Cecchi F, Beani E, Mannari I, Maselli M, Falotico FP, Inguaggiato E, Perazza S, Sicola E, Feys H, Klingels K, Ferrari A, Dario P, Boyd RN, Cioni G. Tele-UPCAT: study protocol of a randomised controlled trial of a home-based Tele-monitored UPper limb Children Action observation Training for participants with unilateral cerebral palsy. BMJ Open. 2018 May 14;8(5):e017819. doi: 10.1136/bmjopen-2017-017819. PMID 29764869
- [Result] Sgandurra G, Biagi L, Fogassi L, Ferrari A, Sicola E, Guzzetta A, Tosetti M, Cioni G. Reorganization of action observation and sensory-motor networks after action observation therapy in children with congenital hemiplegia: A pilot study. Dev Neurobiol. 2020 Sep;80(9-10):351-360. doi: 10.1002/dneu.22783. Epub 2020 Oct 28. PMID 32986904
- [Derived] Ozipek M, Saricaoglu M, Hanoglu L, Mutluay F. Action observation therapy effects on motor function and balance in cerebral palsy: an fNIRS-based randomized trial. Trials. 2025 Nov 3;26(1):465. doi: 10.1186/s13063-025-09181-2. PMID 41184905